CLINICAL TRIAL: NCT01284556
Title: An International, Double-blind, Parallel-group, Placebo-controlled, Randomized Study: Evaluation of the Efficacy and Safety of Phenobarbital as Adjunctive Therapy in Participants (> or = 17 to 70 Years Old) With Partial Onset Seizures
Brief Title: Evaluation Phenobarbital as Adjunctive Therapy in Participants With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West-Ward Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGG-901; 2010-020871-22 (EudraCT Number)
Record Dates: First submitted 2011-01-20; First posted 2011-01-27 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
Keywords: partial onset seizures
MeSH Terms: conditions — Epilepsy | interventions — Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): placebo tablets
  Interventions: Drug: Placebo tablet
- 60 mg group (Experimental): Patients titrated to 60mg phenobarbital for maintenance period, then titrated down.
  Interventions: Drug: Phenobarbital
- 100 mg group (Experimental): Patients titrated to 100mg phenobarbital maintenance period, then titrated down
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: Phenobarbital — tablet
  Arms: 100 mg group; 60 mg group
Drug: Placebo tablet — tablet
  Arms: Placebo

SUMMARY:
Primary:

- to evaluate the efficacy of phenobarbital in reducing seizure frequency.

Secondary:

* to confirm dose response relationship,
* to assess the effects on Type I seizures,
* to assess the safety of phenobarbital
* to assess the drug tolerability.

DETAILED DESCRIPTION:
Primary:

-to evaluate the efficacy of once daily (OD) administration of 60 mg and 100 mg phenobarbital, in reducing seizure frequency in participants with partial onset seizures (Type I seizures; complex or simple with motor symptoms only) not fully controlled despite treatment with 1 to 3 concomitant anti-epileptic drugs (AEDs) or AEDs with Vagus Nerve Stimulator (VNS)

Secondary:

* to confirm dose response relationship of 60 and 100 mg phenobarbital doses,
* to assess the effects of phenobarbital on Type I seizures,
* to assess the safety of phenobarbital
* to assess the tolerability of phenobarbital

ELIGIBILITY:
Inclusion Criteria:

* participants from 17 to 70 years old;
* history of Type I partial onset seizures (complex or simple with motor symptoms only);
* participants must have had electroencephalogram (EEG), magnetic resonance imaging (MRI) or computed tomography (CT) with results consistent with diagnosis of partial-onset seizures;
* participants having at least eight Type I partial onset seizures during 8-week baseline period;
* participants being uncontrolled while treated by 1 to 3 permitted concomitant anti-epileptic drug (AED) and/or Vagus Nerve Stimulation (VNS);
* participant has been on a stable dose of their current anti-epileptic treatment regime

Exclusion Criteria:

* currently taking phenobarbital or primidone;
* currently taking felbamate or vigabatrin;
* history of prior allergic reaction to phenobarbital;
* history of psychogenic seizures;
* history or presence of status epilepticus;
* history or presence of seizures occurring only in clusters;
* participant taking any drug with possible Central Nervous System (CNS) effects except if stable from 1 month prior Visit 1;
* history of cerebrovascular accident (CVA) or transient ischemic attack (TIA);
* presence of any sign suggesting rapidly progressing brain disorder or brain tumor;
* presence of unstable arteriovenous malformations, meningiomas or other benign tumors;
* history of porphyria;
* presence of clinically significant findings on physical exam, vital signs, electrocardiogram (ECG) or safety lab assessments, including renal or hepatic insufficiency;
* history of alcohol or drug abuse within the year prior to screening;
* participant who is known to be non-compliant;
* participant who is male or female who refuses to use an acceptable form of contraception;
* female who is pregnant or lactating or intends to become pregnant;
* participant who has taken part in any investigational device or product within 2 months prior to the screening visit

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of OD administration of 60 mg and 100 mg phenobarbital in reduction of seizure frequency | 34 weeks with maximum 22-week exposure to phenobarbital
  * determination of partial onset seizure frequency per week over the treatment period
  * comparison of average change in weekly seizure rate from baseline and maintenance period

SECONDARY OUTCOMES:
Confirm the dose response relationship of 60 mg and 100 mg phenobarbital doses | 34 weeks with a maximum 22-week exposure to phenobarbital
Assess the effects of phenobarbital on Type I seizures | 34 weeks with a maximum 22-week exposure to phenobarbital
  * seizure freedom rate
  * percent reduction for partial onset seizure
  * responder rate
  * reduction of seizure frequency
Assess the safety of phenobarbital | 34 weeks with a maximum 22-week exposure to phenobarbital
  * overview of adverse events in study
  * summary of adverse events in study by severity, seriousness, relationship to study drug, action taken, outcome, treatment
  * summary of serious adverse events
Assess the tolerability of phenobarbital | 34 weeks with maximum 22-week exposure to phenobarbital

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
- Puerto Rico (2):
  - Hospital Del Maestro, San Juan, PR
  - Centro Neurodiagnostico, Rio Piedras